CLINICAL TRIAL: NCT04606680
Title: Comparative Effectiveness of Herb-partitioned Moxibustion Plus Lifestyle Modification Treatment for Patients With Simple Obesity: A Study Protocol for a Randomized Controlled Trial
Brief Title: Herb-partitioned Moxibustion Plus Lifestyle Modification Treatment for Simple Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hubei Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20201020
Record Dates: First submitted 2020-10-20; First posted 2020-10-28 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Obesity
Keywords: herb-partitioned moxibustion; simple obesity; a randomized controlled trial; effectiveness
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Heat application group (Experimental): Participants will receive heat application at acupoints plus lifestyle modification. Participants will receive heat application treatment once every other day, 3 times per week, for 4 consecutive weeks.
  Interventions: Device: Heat application at acupoints
- Medicated plaster group (Experimental): Participants will receive medicated plaster at acupoints plus lifestyle modification. Participants will receive medicated plaster at acupoints and lifestyle modification every once every other day, 3 times per week, for 4 consecutive weeks.
  Interventions: Device: Medicated plaster at acupoints
- Herb-partitioned moxibustion group (Experimental): Participants will receive herb-partitioned moxibustion at acupoints plus lifestyle modification. Participants will receive herb-partitioned moxibustion at acupoints and lifestyle modification every once every other day, 3 times per week, for 4 consecutive weeks.
  Interventions: Device: Herb-partitioned moxibustion at acupoints

INTERVENTIONS:
Device: Heat application at acupoints — 1. The acupoints will be selected as Tianshu, Pishu, shenshu, zhongwan, and zusanli. The location of the acupoints were based on the national GB/T 12346-2006 acupoints standard. The hot sticker will be placed on the patient's acupoints for about 2 hours. This treatment will be applied once every other day, 3 times per week, for 4 consecutive weeks. The treatment will be delayed during the menstrual period.
  2. The following lifestyle modification are recommended to help to establish healthy habits:
  The proportion of three nutrients in total calories comprises of 55%-65% from carbohydrates, 20%-30% from oils and 15% from protein, and the energy of the whole day distributed to three meals will follow the proportion of 30% for breakfast, 40% for lunch and 30% for dinner. Meanwhile, low-to-moderate intensity physical activities will be instructed to them for at least 5 days per week continually, 30%-50% of the maximum heart rate reserve value will be required.
  Arms: Heat application group
Device: Medicated plaster at acupoints — 1. The acupoints will be selected as Tianshu, Pishu, shenshu, zhongwan, and zusanli. The location of the acupoints were based on the national GB/T 12346-2006 acupoints standard.The chinese traditional medicine(aconite root, dried ginger, evodia rutaecarpa, clove, cinnamon, etc)in moderation will be grinded into powder，and the powder will be added with a certain amount of flour, and finally they will be blended with ginger juice to the appearance of mud. Next, 10g of the kneaded medicine mud will be taked and applied to the bottom of the ordinary sticker. They will be placed on the patient's acupoints for about 2 hours. The sticker has the same shape as the hot sticker, but it does not have the effect of thermal stimulation and infrared radiation. This treatment will be applied once every other day, 3 times per week, for 4 consecutive weeks. The treatment will be delayed during the menstrual period.
  2. Lifestyle modification:It will be performed as the same as the heat application group.
  Arms: Medicated plaster group
Device: Herb-partitioned moxibustion at acupoints — 1. The acupoints will be selected as Tianshu, Pishu, shenshu, zhongwan, and zusanli. The location of the acupoints were based on the national GB/T 12346-2006 acupoints standard[18]. The chinese traditional medicine(aconite root, dried ginger, evodia rutaecarpa, clove, cinnamon, etc)in moderation will be grinded into powder，and the powder will be added with a certain amount of flour, and finally they will be blended with ginger juice to the appearance of mud. Next, 10g of the kneaded medicine mud will be taked and applied to the bottom of the hot sticker. They will be placed on the patient's acupoints for about 2 hours. This treatment will be applied once every other day, 3 times per week, for 4 consecutive weeks. The treatment will be delayed during the menstrual period.
  2. Lifestyle modification:It will be performed as the same as the heat application group.
  Arms: Herb-partitioned moxibustion group

SUMMARY:
This study is designed as a three-dummy randomised controlled trial to evaluate the efficacy and safety of herb-partitioned moxibustion plus lifestyle modification treatment in patients with simple obesity.

DETAILED DESCRIPTION:
This study will be a multicenter, randomized, controlled trial conducted from November, 2018 to November, 2019 that includes 108 participants who have simple obesity and meet the eligibility criteria. The participants will be randomly divided into 3 treatment groups: heat application group, medicated plaster group, or herb-partitioned moxibustion group. Each treatment will last 4 weeks. The primary outcomes will be the clinical effectiveness.The secondary outcome measures include participants'obesity-related indicators, the IWQOL-Lite scale, and the syndrome score of Traditional Chinese Medicine. Adverse events will be recorded during the intervention period.

ELIGIBILITY:
Inclusion Criteria:

Participants meeting all of the following criteria will be considered for inclusion:

1. diagnosed as having simple obesity according to the diagnostic criteria;
2. aged between 18 and 45 years old;
3. Waistline: male≥ 95 cm, women≥85 cm;
4. Being able to fully understand and voluntarily sign informed consent.

Exclusion Criteria:

Participants will be excluded if they have

1. Presence of endocrine disorders such as: polycystic ovary syndrome; Cushing's syndrome; uncorrected thyroid disease.
2. Presence of diabetes mellitus, or hypertension, or abnormal liver and kidney functions, or mental diseases.
3. Pregnant or lactating state, women who plan to become pregnant within 4 weeks.
4. History of bulimia, anorexia, or any other eating disorders.
5. Use of medications in the past 3 months, such as diet drugs, corticosteroids, antidepressants, which may affect weight or appetite.
6. History of surgical weight loss, postoperative adhesions.
7. History of participating in a clinical study of weight loss or any other therapies to lose weight in the past 3 months.
8. Presence of local skin rupture, allergy and scar constitution.
9. Unable to cooperate with the research caused by other diseases or reasons.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Estimated)
Dates: Start 2019-04-30 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
the clinical effectiveness | week 4.
  The clinical effectiveness of 4 weeks of (A)Heat application group, (B)Medicated plaster group, and (C)Herb-partitioned moxibustion group for the improvement of simple obesity will be assessed and determined by the clinical evaluation of nimodipine:
  1. Healing: The clinical symptoms disappear or almost disappear, and the syndrome score is reduced by ≥85 percent;
  2. Significant effect: The clinical symptoms are obviously improved, and the syndrome score is reduced by <85 percent, but ≥50 percent;
  3. Effective: The clinical symptoms have improved, syndrome scores decreased by<50 percent, but ≥30 percent;
  4. Invalid: The clinical symptoms were not improved, even worse, and the syndrome score was reduced by<30 percent.
  Integral variation formula(Nimodipine method: [(pre-treatment score-post-treatment score)/pre-treatment score]X100 percent.

SECONDARY OUTCOMES:
Weight(WG) | week 0, 1, 2, 3, and 4
  Weight(WG) will be measured.
BMI (weight/(height) | week 0, 1, 2, 3, and 4
  BMI (weight/(height) will be measured.
Body fat percentage(F percent) | week 0, 1, 2, 3, and 4
  Body fat percentage(F percent) will be measured.
Waist circumference(WC) | week 0, 1, 2, 3, and 4
  Waist circumference(WC) will be measured.
hip circumference(HC) | week 0, 1, 2, 3, and 4
  hip circumference(HC) will be measured.
waist-to-hip ratio(waist circumference/hip circumference) | week 0, 1, 2, 3, and 4
  waist-to-hip ratio(waist circumference/hip circumference) will be measured.
Visceral fat area | week 0, 1, 2, 3, and 4
  Visceral fat area degree will be measured.
Body fat Obesity degree | week 0, 1, 2, 3, and 4
  Body fat Obesity degree will be measured.
the impact of weight on quality of life (IWQOL)-Lite scale | week 0, 1, 2, 3, and 4
  The impact of weight on quality of life (IWQOL)- Lite scale will be measured. The minimum value is 31，the maximum value is 155. The lower the total score, the lighter the clinical symptoms of the patient.
the syndrome score of Traditional Chinese Medicine | week 0,1,2,3,4.
  The syndrome score of Traditional Chinese Medicine will be adopted as the criterion of syndrome determination according to the diagnostic and therapeutic evaluation standard of simple obesity revised by the 5th National Obesity Research Conference in 1997. The minimum value is 0，the maximum value is 18. The lower the total score, the better of the outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Zhong-Yu Zhou, professor, Principal Investigator — Hubei Hospital of Traditional Chinese Medicine
Locations (1):
- Zhong-Yu Zhou, Hubei, China

REFERENCES:
- [Derived] Wang LH, Lv SY, Liu YR, Chen X, Wang JJ, Huang W, Zhou ZY. Comparative effectiveness of herb-partitioned moxibustion plus lifestyle modification treatment for patients with simple obesity: A study protocol for a randomized controlled trial. Medicine (Baltimore). 2021 Jan 22;100(3):e23758. doi: 10.1097/MD.0000000000023758. PMID 33545941